# Study protocol

**Title:** Impact of a coronary artery calcium-guided primary prevention of major coronary heart disease for asymptomatic coronary artery disease in diabetes: a prospective cohort study

PI: Meng-Huan Lei

CO-PI: Ju-Feng Hsiao, Yu-Chen Hsu

**Affiliations** 

Cardiovascular center, Lo-Tung Poh-Ai Hospital, Taiwan

Version 2, 12/09/2021

# **Background**

The patients with type two diabetes mellites increased gradually and heart disease and cerebral vascular disease is the fourth leading cause of mortality. According to the National Health Insurance Research Database (NHIRD) till 2014, incidence of coronary heart disease is 25.2% and heart failure is 3.77% • Multiple complication including chronic kidney disease and cerebrovascular diseases were also well-known.

A systematic review study of scientific evidence from across the world in 2007-2017 revealed cardiovascular disease (CVD) affected 32.2% overall; 29.1% had atherosclerosis, 21.2% had coronary heart disease (CAD), 14.9% heart failure, 14.6% angina, 10.0% myocardial infarction and 7.6% stroke. CVD representing 50.3% of all deaths is a major cause of mortality among people with type 2 Diabetes mellitus (T2DM) (1).A study in Asian population revealed patients with diabetes had a 1.89-fold risk of all-cause death and 2.0-fold risk of cardiovascular death compared with patients without diabetes(2). However, most diabetes with CAD are asymptomatic.

Coronary artery calcium (CAC) score measured by multi-detector computerized tomography is a reliable measure of subclinical atherosclerosis.

The presence, extent and progression of CAC have been shown to predict adverse cardiovascular events better than traditional risk factors and global risk scoring (3-7) • Our previous study in 2020 revealed CAC score could predict long-term cardiovascular outcomes in asymptomatic patients with T2DM (8). 2019 AHA/ACC Guideline on the Primary Prevention of Cardiovascular Disease and 2019 ESC/EAS Guidelines for the management of dyslipidaemias recommend CAC score as a decision making aid for personalized risk management in primary prevention (9,10). This prospective cohort study will invest the impact of a coronary artery calcium-guided primary prevention of major coronary heart disease for asymptomatic coronary artery disease in T2DM.

## **Objective**

To evaluate benefits of primary prevention of major coronary heart disease for asymptomatic coronary artery disease in T2DM based on the coronary artery calcium score

Our proposal

 Based on CAC score, primary early prevention could reduce incidence of major coronary heart disease (CHD) including cardiac mortality, acute myocardial infarction, coronary revascularization 2.based on CAC score, primary early prevention could reduce all cause mortality, cardiac mortality, cardiovascular disease, heart failure, ischemic stroke, heart failure associated hospitalization and chronic kidney disease and related clinical cost effect.

#### Method

#### Population:

The investigators will enroll 1500 asymptomatic T2DM patients who will receive Coronary artery calcium (CAC) imaging using 256 sliced multidetector computerized tomography (MDCT) scanner as research group and 500 patients as control group from Lan-Yan Diabetes Shared Care Network (public health bureau, clinics, and regional hospital in Yilan County).

Inclusion criteria: more than 40 years old T2DM patients have any one cardiovascular risk as follows

1.total cholesterol > 200mg/dl or low density lipoprotein (LDL) >

- 2.blood pressure > 140/90mm/Hg or taking anti-hypertension agents
- 3.history of smoking
- 4.family history of early coronary heart diseases
- 5.proteinuria

100mg/dl

**Exclusion criteria:** history of cardiovascular diseases such as coronary heart disease, stroke, heart failure etc, pregnant

#### **CAC Scores Measurement**

Coronary artery calcium (CAC) imaging was performed using an 256 sliced multi-detector computerized tomography (MDCT) scanner (Philips Brilliance 256) equipped with high-resolution detectors.

#### Intervention for study group

Based on 2019 AHA/ACC Guideline on the Primary Prevention of
Cardiovascular Disease and 2019 ESC/EAS Guidelines for the management
of dyslipidemias and result of CAC score(9-12), the investigators will
recommend the in-charged doctor to control the cardiovascular risk factors
more aggressively. The study protocols are as follows

If CAC score >0, Treadmill ECG or Thallium<sup>201</sup> Scan would be arranged. If
Treadmill ECG or Thallium<sup>201</sup> show significant ischemia, further study such as
CT angiography or coronary angiography will be arranged.

If CAC score > 100 , Aspirin 100mg QD will be suggested to decrease the cardiovascular risk in patients with low risk of bleeding. Previous studies revealed aspirin for patients with CAC score>100 at low bleeding risk indicated net benefit (13-17).

If CAC score > 400 , statin therapy will be suggested to control lipidemia aggressively and target LDL level < 70 mg/dL (9-12) °

The investigators will follow up these patients every 6 month, record their results of blood tests and medication for 5 years. Primary endpoint is major coronary heart disease including cardiac mortality, acute myocardial infarction and coronary revascularization. Second endpoint include all caused death, death due to cardiovascular disease, heart failure, stroke, admission for heart failure, chronic kidney disease and stroke, and cost related to AMI, coronary heart disease, heart failure, stroke, chronic kidney disease etc.

#### **Control group**

The investigators will enroll 500 age, gender, risk factor matched T2DM patient from our hospital. The doctor in charge will give usual care according to the Diabetes associate of Taiwan clinical practice guidelines for diabetes care.

### Reference

- Einarson TR, Acs A, Ludwig C, Panton UH. Prevalence of cardiovascular disease in type 2 diabetes: a systematic literature review of scientific evidence from across the world in 2007-2017. Cardiovascular diabetology 2018;17:83.
- 2. Yang JJ, Yu D, Wen W et al. Association of Diabetes With All-Cause and Cause-Specific Mortality in Asia: A Pooled Analysis of More Than 1 Million Participants. JAMA network open 2019;2:e192696.
- 3. Dedic A, Ten Kate GJ, Roos CJ et al. Prognostic Value of Coronary Computed Tomography Imaging in Patients at High Risk Without Symptoms of Coronary

- Artery Disease. The American journal of cardiology 2016;117:768-74.
- 4. Raggi P, Shaw LJ, Berman DS, Callister TQ. Prognostic value of coronary artery calcium screening in subjects with and without diabetes. Journal of the American College of Cardiology 2004;43:1663-9.
- 5. Polonsky TS, McClelland RL, Jorgensen NW et al. Coronary artery calcium score and risk classification for coronary heart disease prediction. Jama 2010;303:1610-6.
- 6. Faustino A, Providência R, Mota P et al. Can cardiac computed tomography predict cardiovascular events in asymptomatic type-2 diabetics?: results of a long term follow-up. BMC cardiovascular disorders 2014;14:2.
- 7. Yeboah J, Erbel R, Delaney JC et al. Development of a new diabetes risk prediction tool for incident coronary heart disease events: the Multi-Ethnic Study of Atherosclerosis and the Heinz Nixdorf Recall Study. Atherosclerosis 2014;236:411-7.
- 8. Lei MH, Wu YL, Chung SL, Chen CC, Chen WC, Hsu YC. Coronary Artery Calcium Score Predicts Long-Term Cardiovascular Outcomes in Asymptomatic Patients with Type 2 Diabetes. Journal of atherosclerosis and thrombosis 2021;28:1052-1062.
- 9. Arnett DK, Blumenthal RS, Albert MA et al. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation 2019;140:e596-e646.
- 10. Mach F, Baigent C, Catapano AL et al. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. European heart journal 2020;41:111-188.
- 11. Grundy SM, Stone NJ, Bailey AL et al. 2018

  AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA

  Guideline on the Management of Blood Cholesterol: A Report of the

  American College of Cardiology/American Heart Association Task Force on

  Clinical Practice Guidelines. Circulation 2019;139:e1082-e1143.
- 12. Grundy SM, Stone NJ, Bailey AL et al. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation 2019;139:e1046-e1081.
- 13. Nasir K, Cainzos-Achirica M. Role of coronary artery calcium score in the primary prevention of cardiovascular disease. BMJ (Clinical research ed) 2021;373:n776.

- 14. Ajufo E, Ayers CR, Vigen R et al. Value of Coronary Artery Calcium Scanning in Association With the Net Benefit of Aspirin in Primary Prevention of Atherosclerotic Cardiovascular Disease. JAMA cardiology 2021;6:179-187.
- 15. Cainzos-Achirica M, Greenland P. Coronary Artery Calcium for Personalized Risk Management-A Second Chance for Aspirin in Primary Prevention? JAMA cardiology 2021;6:187-188.
- Cainzos-Achirica M, Miedema MD, McEvoy JW et al. Coronary Artery Calcium for Personalized Allocation of Aspirin in Primary Prevention of Cardiovascular Disease in 2019: The MESA Study (Multi-Ethnic Study of Atherosclerosis). Circulation 2020;141:1541-1553.
- 17. Zheng SL, Roddick AJ. Association of Aspirin Use for Primary Prevention With Cardiovascular Events and Bleeding Events: A Systematic Review and Meta-analysis. Jama 2019;321:277-287.